CLINICAL TRIAL: NCT01277744
Title: A Phase II Study of Hyperthermic Peritoneal Perfusion (HIPEC) for Adolescent and Young Adults With Desmoplastic Small Round Cell Tumor and Other Non-Carcinomas
Brief Title: Pilot Study of Hyperthermic Peritoneal Perfusion (HIPEC) for Adolescent and Young Adults With Desmoplastic Small Round Cell Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0528; NCI-2011-00245 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-01-12; First posted 2011-01-17 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Advanced Cancers; Sarcoma
Keywords: Desmoplastic small round cell tumor; DSRCT; Hyperthermic peritoneal perfusion; HIPEC; Complete abdominal tumor excision; Extensive abdominal disease; Non-carcinoma tumors; Abdominal cavity; Cisplatin; Platinol-AQ; Platinol; CDDP; Diffuse peritoneal tumor; Retroperitoneal tumor; Ovarian germ cell; Wilms' tumor
MeSH Terms: conditions — Sarcoma; Desmoplastic Small Round Cell Tumor; Wilms Tumor | interventions — Hyperthermic Intraperitoneal Chemotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HIPEC + Cisplatin (Experimental): HIPEC, technique for combining hyperthermia and chemotherapeutic agents delivered intraoperatively to the peritoneal and retroperitoneal surface via a recirculating perfusion circuit, performed after cytoreductive surgery and lysis of adhesions. Cisplatin 100 mg/M2 per perfusion catheter. The perfusion is continued for 90 minutes after adding the Cisplatin.
  Interventions: Procedure: Hyperthermic Peritoneal Perfusion (HIPEC); Drug: Cisplatin

INTERVENTIONS:
Procedure: Hyperthermic Peritoneal Perfusion (HIPEC) — HIPEC, technique for combining hyperthermia and chemotherapeutic agents delivered intraoperatively to the peritoneal and retroperitoneal surface via a recirculating perfusion circuit, performed after cytoreductive surgery and lysis of adhesions.
Drug: Cisplatin — 100 mg/M2 per perfusion catheter. The perfusion is continued for 90 minutes after adding the cisplatin.
  Other Names: Platinol-AQ; Platinol; CDDP

SUMMARY:
The goal of this clinical research study is to learn if heated intra-abdominal cisplatin can help to control abdominal tumors in patients having surgery to remove the tumors. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Cisplatin has a platinum atom at its center. The platinum is supposed to poison the cancer cells, which may cause them to die.

Surgery and Study Drug Administration:

If you are found to be eligible, the abdominal surgery will be performed to try to remove as many tumors as possible. The abdominal surgery is not being performed specifically for this research study and would be performed even if you didn't take part in this study. You will be given a separate consent form to sign that explains the details and risks of abdominal surgery in more detail.

During the surgery you will receive sodium thiosulfate by vein. The abdomen will then be temporarily closed. Then the abdominal wash will begin. During the "abdominal wash," heated cisplatin will be delivered through plastic tubing that is connected to a pump into the abdomen. The pump pushes the heated cisplatin into the abdomen and then pulls it out and recirculates the cisplatin. The skin of the abdomen is temporarily closed during the abdominal wash. The surgeon will also "wash" over the closed area of the surgical site. A pump will be used to pump heated cisplatin in and out of the abdomen over 90 minutes while the surgeon gently presses on the abdominal wall so the cisplatin reaches all areas in the abdomen. After 90 minutes, the cisplatin is removed and the abdomen will be "washed" with saline and all fluid will be removed before the surgeon permanently closes the abdomen with 3 layers of stitches.

Two (2) pea-sized tumor samples will be sent to the laboratory of Dr. Dina Lev for tissue evaluation and extraction of RNA (genetic material). One (1) tumor sample will be removed before the procedure and the other sample will be removed at the end of the procedure. The samples will be examined under a microscope and DNA (the genetic material in cells) will be removed to look for any changes to the DNA. The results of these tests will not be shared with you, nor will they be used for any decisions regarding your treatment. The samples will be destroyed after these tests are complete.

There is a chance that the surgeon may decide during the surgery that the abdominal wash will not be performed, for example if the disease has spread to or attached to certain organs. If this occurs, your doctor will discuss other treatment options with you.

Study Visits:

On Days 1-5, 11, and 14, (Day 1 being the day after surgery):

* Blood (about 1 teaspoon) will be drawn for routine tests.
* You will have a physical exam, including measurement of your weight and vital signs.

Follow-Up Visits:

About 1, 3, and 6 months after the surgery is complete, you will have follow-up visits and the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 1 teaspoon) will be drawn at the 1 month visit only for routine tests.
* You will have a hearing test at the 1 month visit only.
* Blood (about 3 teaspoons) will be drawn for routine tests at the 3 and 6 month visits only.
* At the 3 and 6 month visits only, you will have a CT scan, positron emission tomography (PET)-CT scan, or MRI scan to check the status of the disease.

Length of Study:

You will remain on study for up to 6 months. You will be taken off study if the disease gets worse.

If the study doctor learns that the disease has come back or gotten worse at the 6 month follow-up visit, you may be eligible for a re-perfusion, which is a repeat of the operation and study drug administration. If you are eligible for a re-perfusion, your participation on this study will end and then you will be given a new consent form to sign in order to be re-enrolled back onto this study.

This is an investigational study. Cisplatin is FDA-approved and commercially available for the treatment of advanced bladder cancer, metastatic testicular cancer, metastatic ovarian cancer, hepatoblastoma, neuroblastoma, metastatic appendiceal cancer, and abdominal mesothelioma. The use of cisplatin in patients with abdominal sarcoma-type tumors is investigational.

Up to 22 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 1 years
2. Histologically or genetically proven diffuse peritoneal or retroperitoneal tumor from desmoplastic round cell tumor, ovarian germ cell, sarcoma, Wilms' tumor, or other non-carcinoma tumors.
3. Radiologic workup must demonstrate that the disease is confined to the abdominal cavity
4. Radiologic workup or prior abdominal exploration must be consistent with disease which can be debulked to a residual size of less than or equal to 1 cm thickness per tumor deposit
5. Patients must have a minimum expected duration of survival of greater than 6 weeks as determined and documented by the attending surgeon or medical oncologist.
6. Patients must not have any systemic illness which precludes them from being an operative candidate as determined by anesthesia preoperative evaluation. This includes but is not limited to, sepsis, liver failure, pregnant or lactating females.
7. Patients must have fully intact mental status and normal neurologic abilities. Intact mental status is defined by 'the capacity to identify and recall one's identity and place in time and space.' Assessment of mental status and documentation of fully intact mental status will be completed using physical and mental exam by the referring doctor or oncologist.
8. Patients must have adequate renal function (serum creatinine </= 1.5 mg/dl without history dialysis or renal failure or creatinine clearance less than 50 mL/min/1.73M^2 if less than 5 years of age)
9. Patients will be eligible if the white blood cell count (WBC) is >/=2000/microliter or absolute neutrophil count (ANC) is >/=1,500 and platelets are >/= 100,000/mm^3
10. Patients will be eligible if serum total bilirubin and liver enzymes are </=2 times the upper limit of normal
11. Patients must be recovered from any toxicity from all prior chemotherapy, immunotherapy, or radiotherapy and be at least 14 days past the date of their last treatment

Exclusion Criteria:

1. Patients will be ineligible if they have any concomitant cardiopulmonary disease which would place them at unacceptable risk for a major surgical procedure
2. Patients will be ineligible if they have disease outside of the abdominal cavity which is uncontrolled
3. Patients will be ineligible if they have a baseline neurologic toxicity of Grade 3 or greater (because of the potential neurotoxicity associated with platinum)
4. Patients who have failed previous intraperitoneal platinum therapy will be ineligible
5. Patients with Retroperitoneal Liposarcoma will be ineligible.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-05-09 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hayes-Jordan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.utmdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details: May 2011 to December 2013
Pre-assignment Details: One patient was enrolled twice; she received a second hyperthermic intraperitoneal chemotherapy surgery after she recurred following the first procedure
Groups:
- HIPEC: HIPEC with Cisplatin
Period: Overall Study
Arm/Group | HIPEC
Started | 22
Completed | 20
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | HIPEC
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 21
  Russia | 1

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival
Description: Date of surgery to date of death or date of recurrence, whichever occurred first for patients who experienced an event, and to date of last follow-up for patients alive without recurrence
Time Frame: 36 months after the last participant enrolled
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HIPEC
Number analyzed (Participants) | 20
months | 13.99 [7.26 to NA] — 95 percent are upper limit was not estimable

2. Secondary Outcome: Overall Survival
Description: From the date of diagnosis to the date of death or last follow up date for patient alive.
Time Frame: From the date of diagnosis to the date of death or last follow up date for patient alive up to 81 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HIPEC
Number analyzed (Participants) | 20
months | 58.4 [43.7 to NA] — 95 percent are upper limit was not estimable

ADVERSE EVENTS:
Time Frame: 6 months post surgery
Arm/Group | HIPEC
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 18/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIPEC (N=20)
Creatinine increased (Investigations) | 2
White blood cell decreased (Investigations) | 14
Platelet count decreased (Investigations) | 15
Neurogenic bladder (Gastrointestinal disorders) | 3
Urinary tract infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT01277744/Prot_SAP_000.pdf